CLINICAL TRIAL: NCT01398631
Title: A Prospective Comparison of the TIMI, GRACE and HEART Scores for Predicting Cardiovascular Events in Chest Pain Patients in the Emergency Room
Brief Title: A Comparison of the TIMI, GRACE and HEART Scores
Acronym: HEART
Status: Completed | Type: Observational
Sponsor: R&D Cardiologie (Other)
Collaborators: Sanofi (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, Barbra Backus, MD, PhD, R&D Cardiologie
Other Study IDs: Z-08.27
Record Dates: First submitted 2010-06-09; First posted 2011-07-20 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Risk scores; ACS; HEART-score
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: All included patients presented with chest pain at the emergency room within the inclusion period.

SUMMARY:
Various elements of patient history are checked and entered in the admission Case Recor Form (CRF). Three risk scores are calculated out of these elements, combined with physical examination, laboratory values and ECG-findings.

The primary aim is to assess the positive and negative predictive values for a cardiovascular event of the three risk scores for chest pain patients.

Secondary aim is to assess the sensitivity and specificity of various elements in the patient history for an acute coronary syndrome.

DETAILED DESCRIPTION:
This is a prospective, observational study in patients admitted to the emergency room for chest pain. All patients are checked by the resident in charge immediately on admission, before any lab values are known, by means of an admission Case Report Form (CRF), consisting of classical elements of patient history, risk factors, medication and physical examination. This CRF is filled out immediately by the resident. No additional effort will be asked of the patients.

Patient data during a follow up of at least 6 weeks are gathered from hospital charts.

The predictive value of the three scoring systems: HEART (History, ECG, Age, Risk factors, Troponin), TIMI (Thrombolysis in Myocardial Infarction) and GRACE (Global Registry of Acute Coronary Events) for both the discharge diagnosis and the occurrence of Major Adverse Cardiovascular Events (MACE) is calculated.

The primary hypothesis of the study is that the HEART score is a significantly better predictor than the TIMI and/or GRACE score for cardiovascular events during a six week period following admission to the emergency room.

ELIGIBILITY:
Inclusion Criteria:

* any patient visiting the cardiology emergency room due to chest pain

Exclusion Criteria:

* chest pain clearly due to rhythm disturbances or acute heart failure
* concomitant non cardiac disease with expected fatal outcome within 1 year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presentating with chest pain in one of the participating hospitals.
Sampling Method: Probability Sample
Enrollment: 2440 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Occurence of MACE (Major Adverse Cardiac Events) | 6 weeks after presentation
  The number of patients diagnosed with MACE (Acute Myocardial Infarction, Percutaneous Coronary Intervention, Coronary Artery Bypass Grafting, Significant stenosis with conservative therapy, Death)

SECONDARY OUTCOMES:
The number of patients undergoing Coronary ArterioGraphy (CAG) | Three months after presentation
The number of patients suffering Acute Coronary Syndrome (ACS) | 3 months after presentation
  According to adjudication committee

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Doevendans, MD,PhD,Prof, Study Chair — UMC Utrecht; Barbra Backus, MD, Principal Investigator — St Antionius Hospital Nieuwegein; Jacob Six, MD, PhD, Study Director — Hofpoort Hospital Woerden
Locations (10):
- Netherlands (10):
  - Meander Medical Centre, Amersfoort
  - Gelre Hospital, Apeldoorn
  - Reinier de Graaf Gasthuis, Delft
  - University Medical Centre Groningen, Groningen
  - Medical Centrum Haaglanden, Leidschendam
  - St Antonius Hospital, Nieuwegein
  - Medical Centre Haaglanden, The Hague
  - St Antonius Hospital, Utrecht
  - University Medical Centre Utrecht, Utrecht
  - Hofpoort Hospital, Woerden